CLINICAL TRIAL: NCT04639388
Title: Characterize the Behavioral Prodromes of Psychotic Disorders in Children With 22q11.2DS Aged From 4 to 13 Years Old
Brief Title: Understanding of Psychotic Disorders in Children With 22q11.2DS
Acronym: PremiCeS22
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A01370-39
Record Dates: First submitted 2020-10-01; First posted 2020-11-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: 22q11.2 Deletion Syndrome
MeSH Terms: conditions — DiGeorge Syndrome | interventions — Neuropsychological Tests; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Monocentric study with two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22q11.2DS (Experimental): Children aged from 4 to 13 years old with 22q11.2 deletion syndrome
  Interventions: Behavioral: neuropsychological testing, questionnaires and experimental tasks
- Control Group (Non22q11.2DS) (Active Comparator): Children aged from 4 to 13 years old without developmental disease
  Interventions: Behavioral: neuropsychological testing, questionnaires and experimental tasks

INTERVENTIONS:
Behavioral: neuropsychological testing, questionnaires and experimental tasks — Neuropsychological testing (the Sky Search subtest from the Test of Everyday Attention for Children (TEA-Ch); the Overlapping lines task of Rey; auditory attention of NEPSY II battery); questionnaires completed by the children's legal representatives to assess behavior; experimental tasks evaluating gaze direction and facial expression recognition

SUMMARY:
The study PremiCeS22 will investigate the prodromal signals at the onset of psychotic disorders of children with 22q11.2 deletion syndrome

DETAILED DESCRIPTION:
22q11.2DS is one of the most common microdeletion syndromes (1 / 2000-1 / 4000 births) and one of the most robust genetic risk factors for schizophrenia (1 to 2% of cases). Reciprocally, approximately 30% of patients with 22q11.2DS will develop psychotic symptoms in adolescence or early adulthood. It is now well established that children and adults with 22q11.2DS have lower social skills than developing youth. These social dysfunctions could be partly underpinned by alterations in social cognitive processes, and could also be linked to the emergence of psychotic signs or even schizophrenia. However, to our knowledge, no study has investigated the existence of behavioral prodromal signs during the onset of psychotic signs in children with 22q11.2DS. In addition, the origin of social cognitive processes remains to this day little explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 22q11.2 deletion syndrome or no developmental disease
* Aged from 4 to 13 years old
* French language

Exclusion Criteria:

* Diagnosis of intellectual deficiency according to DSM 5 criteria
* Drug prescribed for somatic condition that could influence cerebral functioning

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The Screen for child Anxiety Related Emotional Disorders (SCARED) | Day 1
  Scale assessing behavioral prodromes or warning signs of hallucinations in psychotic disorders A psychometric study is then carried out on this questionnaire in order to validate it with parents of children carrying 22q11.2DS.
facial expression recognition task | Day 1
  Proportion of correct responses in experimental tasks evaluating gaze direction and facial expression recognition

SECONDARY OUTCOMES:
Sustained hearing attention test (Tea-Ch battery) | Day 1
  Proportion of impaired scaled score at the Sky Search subtest from the Test of Everyday Attention for Children (TEA-Ch)
Rey's Tangled Lines Test | Day 1
  Proportion of impaired scaled score to study the degree of cognitive development in children
NEPSY II battery | Day 1
  Proportion of impaired scaled score at auditory attention of NEPSY II battery The NEPSY-II is a comprehensive neuropsychological battery for children ages 3-12. The test provides measures of sensor-motor, language, visuospatial processing, memory and learning, attention/executive functions, and social cognition.
Mean reaction time | Day 1
  Mean reaction time in neuropsychological testing and experimental tasks

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noëlle BABINET, Principal Investigator — CH LE VINATIER
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No